CLINICAL TRIAL: NCT05604365
Title: FearLess in Cognitively Intact Patients With Glioma
Acronym: FearLess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-22-19485; HM20025081 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2022-10-26; First posted 2022-11-03 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Glioma; Fear of Cancer
MeSH Terms: conditions — Glioma; Pathophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Patients Only
  Interventions: Behavioral: FearLess Intervention
- Arm 2 (Experimental): Patients and Caregivers
  Interventions: Behavioral: FearLess Intervention
- Arm 3 (Experimental): Caregivers Only
  Interventions: Behavioral: FearLess Intervention

INTERVENTIONS:
Behavioral: FearLess Intervention — 8-12 weekly telehealth sessions one hour in length.The intervention includes psychotherapy techniques varying from relaxation response to self-regulation targeted to the specific fears of patients with glioma.

SUMMARY:
This study will assess the preliminary feasibility and acceptability of FearLess, a newly-developed psychological intervention for fear of cancer recurrence (FCR) among cognitively-intact patients with glioma.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion:

* Confirmed glioma diagnosis (grade II-IV) via histopathology
* Be a minimum of 2 weeks post surgical repair or biopsy (if applicable)
* Elevated FCR [> 13 on Fear of Cancer Recurrence Inventory]
* Primarily English speaking

Caregiver Inclusion:

* Loved one, or non-paid care partner to a patient with a confirmed glioma diagnosis (grade II-IV) via histopathology
* Elevated FCR [> 13 on Fear of Cancer Recurrence Inventory]
* Primarily English speaking
* Age 18+

Exclusion Criteria:

Patient:

* Cognitive impairment [< or equal to 31 on the Telephone Interview for Cognitive Status (TICS)]
* Inability to attend virtual sessions (e.g. due to lack of stable internet connection, difficulty using technology)
* Inability to understand and provide informed consent.

Caregiver:

* Inability to attend virtual sessions (e.g. due to lack of stable internet connection, difficulty using technology)
* Inability to understand and provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Determine feasibility of FearLess recruitment | 1 Day
  As evidenced by the number of patients and caregivers that enroll in the trial
Determine the feasibility of FearLess intervention- Data collection procedures | 12 Weeks
  As evidenced by the number of participants that complete the baseline assessment, post-intervention assessment, and the exit interview
Determine the acceptability of FearLess intervention- Attendance | 12 Weeks
  As evidenced by attendance rate at intervention sessions
Determine the acceptability of FearLess intervention- Retention Rate | 12 Weeks
  As evidenced by the number of patients that complete follow-up measures
Determine the acceptability of FearLess intervention- Satisfaction | 12 Weeks
  As evidenced by the number of patients with a satisfaction rating greater than 7 on a 10 point scale
Determine the acceptability of FearLess intervention- Satisfaction- Recommendation | 12 Weeks
  As evidenced by the number of patients that recommend the intervention to others

OTHER OUTCOMES:
Determine the efficacy of FearLess intervention- Baseline to post intervention - fear scale | 12 Weeks
  As determined by the number of patients and caregivers that demonstrate meaningful reductions in self-reported fear of cancer recurrence, utilizing a 49 item scale assessing fear of cancer recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Ashlee Loughan, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT05604365/ICF_000.pdf